CLINICAL TRIAL: NCT05428800
Title: The Effect of Progressive Relaxation Exercises on Premenstrual Syndrome Symptoms: Randomized Controlled Study
Brief Title: The Effect of Progressive Relaxation Exercises on Premenstrual Syndrome Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Elif TUGCE CITIL, Assistant professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-41997688-050.99-43313
Record Dates: First submitted 2022-06-09; First posted 2022-06-23 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual Syndrome, Exercises, Women Health
MeSH Terms: conditions — Premenstrual Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Progressive relaxation exercises will be performed for 25-30 minutes every day for 8 weeks, and at the end of 8 weeks, the group will be evaluated again with PMSS.
  Interventions: Behavioral: Progressive Relaxation Exercises
- Control (No Intervention): They will continue their routine coping habits for 8 weeks, and at the end of 8 weeks, the group will be evaluated again with PMSS.

INTERVENTIONS:
Behavioral: Progressive Relaxation Exercises — Progressive muscle relaxation (PMR) is a relaxation technique that tenses and relaxes muscles in an unprompted, regular, and consecutive manner until the whole body is relaxed.
  Arms: Experimental

SUMMARY:
The aim of this study; to determine the effect of progressive relaxation exercises on premenstrual syndrome symptoms. The study is a randomized controlled trial, and women between the ages of 18-35 who meet the inclusion criteria will be included. Participant information form and premenstrual syndrome scale will be used in the research. There are two groups in the study as experimental (n=40) and control (n=40).

DETAILED DESCRIPTION:
Institutional permission and ethics committee approval were obtained for the research. The population of the study consisted of 218 women. The sample of the study consisted of 80 women, 40 of which were experimental and 40 control. Participants were evaluated according to the www.randomizer.org program and randomization was achieved among the women participating in the study.

The research process and the participants in the experimental and control groups will be explained again and the necessary equipment will be provided by the researchers. The "Progressive Relaxation Exercises Guide" prepared by the researcher in accordance with the literature will be given to the women in the experimental group (40), taking the opinions and suggestions of eight experts. At the same time, the comprehensibility and applicability of the guide were evaluated by making a pilot application to 10 women before the research. Afterwards, all the information in the guide will be explained to the women in the experimental group and training will be given until adequate feedback is received. At the same time, progressive relaxation exercises belonging to the Turkish Psychological Association were given to the women in CD form, and listening to the audio recordings together with the relaxation exercises to be performed in accordance with the guide will be indicated. These exercises will be performed by the women in the experimental group for 25-30 minutes a day, every day for 8 weeks. At the end of 8 weeks, women will be reassessed with PMSS. The women in the control group (40) will be told to continue their routine habits regarding PMS in parallel with the study group, without any application. At the end of 8 weeks, women in the control group will be re-evaluated with PMSS.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-35 years old, single marital status,
* Willingness and volunteering to work,
* Being able to read and write in Turkish and understand what he reads,
* Applying to the obstetrics and gynecology outpatient clinic for routine control,
* Getting a score of 110 and above in PMSS.

Exclusion Criteria:

* The woman has an obstetric or medical health problem that prevents her from doing progressive relaxation exercises,
* Having a chronic and gynecological health problem,
* Regular exercise,
* There is a change in menstrual characteristics in the last six months.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The research was conducted with women between the ages of 18-35.
Enrollment: 79 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
intervention applied to the experimental group | It includes an 8-week process.
  At the end of 8 weeks of progressive relaxation exercises, improvement in premenstrual syndrome symptoms of the experimental group is expected.

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Science University, Kütahya, Turkey (Türkiye)